CLINICAL TRIAL: NCT03290625
Title: Intranasal Sedation With Dexmedetomidine and Ketamine in Pediatric Dentistry (NASO II): Randomized Clinical Trial
Brief Title: Intranasal Sedation With Dexmedetomidine and Ketamine in Pediatric Dentistry (NASO II)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de Goiás (FAPEG) (Unknown)
Responsible Party: Principal Investigator, Luciane Ribeiro de Rezende Sucasas da Costa, Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PV0939-2017
Record Dates: First submitted 2017-09-14; First posted 2017-09-25 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Caries of Infancy; Dental Anxiety
MeSH Terms: interventions — Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DexKet (Experimental): Intranasal DEXMEDETOMIDINE (2.0 mcg/kg, maximum 100 mcg) + KETAMINE (1.0 mg/kg, maximum 100 mg)
  Interventions: Drug: Dexmedetomidine Hydrochloride; Drug: Ketamine Hydrochloride
- Dex (Active Comparator): DEXMEDETOMIDINE (2.5 mcg/kg, maximum 100 mcg)
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Dexmedetomidine hydrochloride (PrecedexTM), presented in ampoule containing 2 mL of 100 mcg / mL solution for injection
Drug: Ketamine Hydrochloride — Dextrocetamine hydrochloride (KetaminTM), presented in a 10 mL vial containing 50 mg / mL solution for injection
  Arms: DexKet

SUMMARY:
Parallel clinical trial focusing on procedural pediatric sedation in the dental setting. Children will be randomized to treatment according to a predetermined sequence of interventions consisting of: 1. intranasal sedation with ketamine-associated dexmedetomidine (Experimental Group), 2. intranasal sedation with dexmedetomidine as sole drug (Control Group). Primary outcome is children's behavior during the dental treatment. Secondary outcomes are: children's pain, memory and stress (salivary cortisol and melatonin); perception of the accompanying adult, dentist and child about dental sedation; cost-effectiveness of this type of sedation; psychosocial variables; children's quality of life.

DETAILED DESCRIPTION:
This proposal aims to determine the most effective pharmacological regimen in the treatment of child pain and anxiety during outpatient dental procedures. Advancement in this field is a reflection, on the one hand, of the use of new and more effective routes of drug administration, such as the intranasal route using atomizers with uniform dispersion of the administered jet and, on the other hand, the use of new sedative drugs, such as dexmedetomidine. This is a randomized, parallel, triple-masked clinical trial, using a research protocol with the objectives: 1) To evaluate the efficacy (behavior, pain, memory and stress) of a sedative regimen intranasally mucosal atomizer device (MAD) using a sedative drug (ketamine) and an innovative drug (dexmedetomidine) in the sedation of children from 2 to 6 years of age undergoing dental treatment - our hypothesis is that the use of dexmedetomidine intranasally association with ketamine is more effective than dexmedetomidine itself in isolation; 2) To analyze the level of cortisol and salivary melatonin (stress) according to each sedative protocol and its association with clinical variables; 3) Identify adverse events with the new protocol; 4) To evaluate the association between the child's behavior and psychosocial variables; 5) To verify the impact of treatment under dental sedation on the quality of life related to the oral health of the child. The research will be carried out in the Faculty of Dentistry of the Federal University of Goias, in the Center of Studies in Dental Sedation (NESO), Goiânia, Goias. A non-probabilistic sample of 88 children aged 2 to 6 years (alpha 0.05, 80% power) who present dental caries with restorative need, American Society of Anesthesiologists I or II, patent nasal airways (Mallampati index I or II and obstruction by hypertrophy of tonsils ≤ 50% and effective nasal breathing), in addition to non-cooperative behavior with the examination or a dental procedure. Children with neuropathies, those using growth hormone and / or those who exhibit severe adverse events during sedation will be excluded. Children will be randomized to treatment according to a predetermined sequence of interventions consisting of: 1. intranasal sedation with ketamine-associated dexmedetomidine (Experimental Group), 2. intranasal sedation with dexmedetomidine as sole drug (Control Group). Pediatricians and anesthesiologists will be aware of the randomized intervention, because of safety concerns for the child, in the case of serious adverse events with or without immediate use of antagonists; the other staff members and the child's companion (s) will be "masked". The examination and intervention sessions will be filmed in high definition for later analysis of the behavior and pain according to different scales consecrated and / or validated. In addition, the children will be submitted to four saliva collections to analyze the levels of cortisol and melatonin (stress-related hormones). Other variables of secondary outcome are: perception of the accompanying adult, dentist and child about dental sedation and cost-effectiveness of this type of sedation, psychosocial variables, quality of life. The data will be analyzed by descriptive and bivariate statistics. This proposal will bring benefits in the vast field of health sedation by having original design, using drugs and promising routes, with national and international impact. The project is inserted in a research line that presents experience history and impact publications by the proponent team, as well as involving students of scientific initiation, master's, doctorate, and postdoctoral studies, being developed by a multidisciplinary team. There is a clear expectation of generating results with high impact production, besides the possibility of immediate application in the public and private sectors of a highly effective sedative regime, minimizing the need to refer patients to general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Children born to term, whose physical condition is categorized as American Society of Anesthesiologists I (healthy) or II (mild and controlled systemic disease - persistent asthma, for example)
* Children with a low risk of airway obstruction (Mallampati less than 2 and / or tonsil hypertrophy occupying less than 50% of the oropharynx)
* Children without neurological or cognitive alterations and who do not use medications that may compromise cognitive functions
* Children with caries requiring dental restoration

Exclusion Criteria:

* Children with positive behavior in the consultation without sedation
* Children with facial deformity
* Children using corticosteroid

Ages: 20 Months to 83 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Children's behavior according to observational scale | From the beginning to the end of the dental treatment, which should last around 30-40 minutes
  Children's behavior during the dental treatment under sedation according to the observational scale 'Ohio State University Behavioral Rating Scale' (OSUBRS) as assessed by trained and calibrated observers in the video files of the procedure

SECONDARY OUTCOMES:
Acceptance of intranasal administration according to observation | From the beginning to the end of the intranasal sedative administration, which should less than one minute each
  Acceptance of intranasal sedative regimen administration using a pre-defined form; trained and calibrated observers will assess children's acceptance through symptoms such as crying, need for physical restraint, and others
Memory of the procedure through questionnaire | From the children's arrival at the dental clinic until discharge, and then on the day after, up to 36 hours
  Children's memory of facts that happened just before and after the administration of the sedative, through a questionnaire exploring toys showed and procedures occurred just before and during the procedure
Salivary cortisol according to ELISA | From the night before the procedure until the end of the dental procedure under sedation, up to 24 hours
  Children's salivary cortisol related to the dental treatment under sedation assessed through ELISA
Salivary melatonin according to ELISA | From the night before the procedure until the end of the dental procedure under sedation, up to 24 hours
  Children's salivary melatonin related to the dental treatment under sedation assessed through ELISA
Pain according to the FLACC scale | From the beginning to the end of the dental treatment, which should last around 30-40 minutes
  Children's pain during the dental treatment under sedation, assessed by trained and calibrated observers using the Faces, Legas, Activity, Consolability and Crying scale (FLACC) in digital video files related to the procedure
Accompanying person perception through VAS | Just after the end of the child's dental procedure, while in the recovery anesthetic room, an average of 60 minutes
  Accompanying person perception on the child's sedation through Visual Analogue Scale
Pediatric dentist perception through VAS | Just after the end of the child's dental procedure, an average of 60 minutes
  Pediatric dentist perception on the child's sedation through Visual Analogue Scale
Child's perception through qualitative interview | One week after the dental sedation procedure
  Child's perception on the dental procedure under sedation, according to a qualitative interview following a semistructured guide
Adverse events | During the procedure and within the 24 hours after
  Post-operative adverse events related to the dental sedation procedure
Child's dental anxiety and sedation efficacy, according to the Venham's picture test | Fifteen minutes before the administration of the sedative
  Association of child's dental anxiety with the outcome of the procedural sedation, using the Venham Picture Test
Child's dental behavior in the reception and sedation efficacy, according to the Sharath Scale | Fifteen minutes before the administration of the sedative
  Association of child's dental behavior with the outcome of the procedural sedation, using the Sharath scale
Parents' anxiety and sedation efficacy, according to the STAI | On the day of the inclusion of the child in the RCT, an average of 30 minutes before the child's dental exam
  Association of parental overall anxiety with the outcome of the procedural sedation, using short form of the State-Trate Anxiety Inventory (STAI)
Parents' dental anxiety and sedation efficacy, according to the Corah Scale | On the day of the inclusion of the child in the RCT, an average of 30 minutes before the child's dental exam
  Association of parental dental anxiety with the outcome of the procedural sedation, using Dental Anxiety Scale by Corah
Parents' overall stress and sedation efficacy, according to the Lipp Inventory | On the day of the inclusion of the child in the RCT, an average of 30 minutes before the child's dental exam
  Association of parental stress with the outcome of the procedural sedation, using the according to the "Inventário de Sintomas de Stress para Adultos de Lipp - ISSL" (Lipp Adult Stress Symptoms Inventory - ISSL)
Procedural dental sedation impact according to the B-ECOHIS | Two weeks and three months after the completion of the dental treatment
  Impact of dental treatment under sedation on the oral health related quality of life related to the child and respective family, using the questionnaire B-ECOHIS
Economic analysis | After the completion of data collection for the primary outcome, an average of 4 years
  Cost-effectiveness analysis of the two sedative regimens

CONTACTS AND LOCATIONS:
Overall Officials: Luciane Costa, PhD, Principal Investigator — Universidade Federal de Goias
Locations (1):
- Dental School, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Undecided